CLINICAL TRIAL: NCT00422487
Title: Phase 2a, Randomized, Double-Blind, Placebo-Controlled Multiple Ascending Dose Study of MBX-2044 to Evaluate the Multiple-dose Pharmacokinetics, Safety and Tolerability When Administered Orally in Patients With Type 2 Diabetes
Brief Title: Safety and Tolerability Study of MBX-2044 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M2044-20610
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- MBX-2044 1.5 mg (Experimental)
  Interventions: Drug: MBX-2044
- MBX-2044 4.5 mg (Experimental)
  Interventions: Drug: MBX-2044
- MBX-2044 15 mg (Experimental)
  Interventions: Drug: MBX-2044
- MBX-2044 30 mg (Experimental)
  Interventions: Drug: MBX-2044
- MBX-2044 60 mg (Experimental)
  Interventions: Drug: MBX-2044
- MBX-2044 90 mg (Experimental)
  Interventions: Drug: MBX-2044
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo for MBX-2044

INTERVENTIONS:
Drug: MBX-2044 — MBX-2044 1.5 mg one capsule daily for 14 days
  Arms: MBX-2044 1.5 mg
Drug: MBX-2044 — MBX-2044 4.5 mg three 1.5 mg capsules daily for 14 days
  Arms: MBX-2044 4.5 mg
Drug: MBX-2044 — MBX-2044 15 mg one capsule daily for 14 days
  Arms: MBX-2044 15 mg
Drug: MBX-2044 — MBX-2044 30 mg two 15 mg capsules daily for 14 days
  Arms: MBX-2044 30 mg
Drug: MBX-2044 — MBX-2044 60 mg one capsule daily for 14 days
  Arms: MBX-2044 60 mg
Drug: MBX-2044 — MBX-2044 90 mg one 60 mg capsule and two 15 mg capsules daily for 14 days
  Arms: MBX-2044 90 mg
Drug: Placebo for MBX-2044 — Placebo Intervention
  Arms: Placebo

SUMMARY:
The purpose of this study is to collect important information regarding the glucose-lowering efficacy of MBX-2044 and the safety of MBX-2044 (especially weight gain and edema) in diabetics. It will also provide important information about the appropriate doses to be used in subsequent longer-term studies to evaluate the safety and efficacy of MBX-2044 alone and in combination with other anti-diabetic agents.

DETAILED DESCRIPTION:
The current study is designed to test the short-term effectiveness and tolerability of MBX-2044 in patients with type 2 diabetes who are currently being controlled with up to one or two non-TZD hypoglycemic agent(s) including sulfonylureas, meglitinides, metformin, α-glucosidase inhibitors or Byetta®. Eligible patients will be enrolled into one of the following treatment cohorts receiving either placebo or MBX-2044 at 1.5, 4.5, 15, 30, or 60 mg/day in a double-blinded study for a 14-day treatment period. Patients will be evaluated for adverse events and vital signs daily. All efficacy and laboratory safety measures will be assessed after 2 weeks. This study will provide important information regarding the glucose-lowering efficacy of MBX-2044 and the safety of MBX-2044 (especially weight gain and edema) in diabetics. It will also provide important information about the appropriate doses to be used in subsequent longer-term studies to evaluate the safety and efficacy of MBX-2044 alone and in combination with other anti-diabetic agents.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes previously controlled with up to one or two non-TZD hypoglycemic agents including sulfonylureas (e.g., glyburide, glipizide, glimeprimide), meglitinides (e.g., Prandin®, Starlix®), metformin (e.g., Glucophage®), α-glucosidase inhibitors (e.g.,acarbose, miglitol) or Byetta®
* All female patients must be either surgically sterile or post-menopausal.
* Male patients with female partners of childbearing potential must agree to use condoms, or their partner must use a medically acceptable form of contraception.
* BMI 24-44 kg/m2.
* Patients must have a FPG ≤ 200 mg/dL at screening.
* Patients must have Hemoglobin A1c ≥ 6.5%, ≤ 10.0% at screening.
* Electrocardiogram (ECG) and chest x-ray must be normal, or considered not clinically significant, for participation in this study.
* Patients must have a blood pressure ≤ 160/90 mm/hg including hypertensive patients controlled with medication.

Exclusion Criteria:

* History of Type 1 diabetes or diabetes secondary to pancreatitis or pancreatectomy.
* History of TZD use (Actos or Avandia) within 6 months of Screening Visit.
* History of TZD discontinuation due to lack of efficacy.
* History of congestive heart failure within last 5 years.
* History of significant pulmonary disease, myocardial infarction, cerebrovascular accident, or nephrotic syndrome within last 1 year.
* Malignancy within the last 5 years (except resected basal cell carcinoma).
* Ongoing active infection.
* Change in treatment with lipid-lowering agent within 7 days of screening visit.
* Current or expected requirement for anticoagulant therapy [except for low-dose aspirin ≤ 325 mg/d or Plavix® ≤ 75 mg/d].
* Current or expected treatment with phenytoin for the duration of the study.
* Known hypersensitivity to NSAIDs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the multiple-dose pharmacokinetics of MBX-2044 administered as monotherapy at the protocol-specified daily dose orally for 14 days
Evaluate the clinical safety and tolerability of MBX-2044 after 14 days administration, including the parameters of weight gain and edema
Determine the maximum tolerated dose (MTD) of MBX-2044, after 14 days administration
Determine the effect of MBX-2044 after 14 days administration, on efficacy parameters

CONTACTS AND LOCATIONS:
Overall Officials: Sherwyn Schwartz, MD, Principal Investigator — Diabetes and Glandular Research Associates
Locations (1):
- Diabetes and Glandular Disease Research Associates, San Antonio, Texas, United States